CLINICAL TRIAL: NCT00285610
Title: Early Exposure to Lead and Adult Antisocial Outcomes
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11261-CP-003
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Lead Poisoning
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Prior research indicates a link between early lead exposure and risk for delinquent behavior. In this study, we follow a large birth cohort from the Cincinnati Lead Study into early adulthood to determine whether this increased risk persists. Outcome measures include official arrest records, diagnoses of Substance Abuse Disorder and Antisocial Personality Disorder, self-report of delinquent behavior, and a psychopathy scale. Predictors include pre-natal and post-natal blood lead levels. Multivariate statistical methods will control for potential confounders/covariates.

ELIGIBILITY:
Inclusion Criteria: (1) Part of original CLS birth cohort -

Exclusion Criteria: (1) Moved out of geographic area

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women were recruited from four prenatal clinics in Cincinnati, Ohio if they resided in areas of the city with a high concentration of older, lead-contaminated housing
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2001-11; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Lead Exposure and Antisocial Behavior | Prenatal (1-2 trimester) and postnatal on a quarterly and bi-annual basis (until 6.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: M. Douglas Ris, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center, Cincinnati, Ohio, United States